CLINICAL TRIAL: NCT03189134
Title: Utilization of Confocal Microscopy During Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aditya Kaza (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Aditya Kaza, Associate in Cardiac Surgery, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P00013570; R56HL128813 (NIH)
Record Dates: First submitted 2017-05-22; First posted 2017-06-16 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial | interventions — Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Imaging arm (Experimental): Up to 5mL of 1:1000 dilute FLUORESCITE will be applied to cardiac tissue prior to imaging with Cellvizio 100 Series System with Confocal Miniprobes
  Interventions: Drug: Fluorescite; Device: Cellvizio 100 Series System with Confocal Miniprobes

INTERVENTIONS:
Drug: Fluorescite — Dilute fluorescite will be applied to cardiac tissue prior to imaging
  Other Names: fluorescein sodium
Device: Cellvizio 100 Series System with Confocal Miniprobes — Microscopy system will image cardiac tissue.

SUMMARY:
The investigators propose to translate confocal microscopy for use during open heart surgery. This tool will help discriminate between various types of tissues in the heart during surgery. One of the most feared complication after heart surgery is heart block. This flexible fiberoptic confocal microscope will help discriminate between the various types of tissues in the heart and thus help avoid injury to the conduction tissue during surgery.

DETAILED DESCRIPTION:
This is an interventional pilot study that proposes to evaluate the safety, logistical feasibility, and technological feasibility of using Fluorescite with fiberoptic confocal microscopy during cardiac surgery to discriminate between cardiac tissue and conduction tissue. During surgery to repair atrial septal defect, diluted Fluorescite will be added to the surface of the heart. The fiberoptic confocal microscope (Cellvizio 100 Series System with Confocal Miniprobe) will be used to record images in several different locations of the heart. The image files will be provided to blinded raters who will attempt to identify whether they contain cardiac tissue or conduction tissue. All subjects will be monitored while they are inpatient after surgery for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 30 days and 21 years old
* Undergoing elective surgery for closure of atrial septal defect
* Both parents attend pre-operative clinic appointment, to provide 2 parent consent, or an adult participant (age 18-21) may provide consent for him/herself

Exclusion Criteria:

* Prior history of adverse reaction to fluorescein sodium
* Prior history of renal failure or abnormal renal function
* Baseline PR interval > 220 msec or 98% for age
* Baseline HR > 87% for age
* Underlying genetic syndrome associated with progressive AV block of sinus node dysfunction (e.g. Holt-Oram or NKX2.5)

Ages: 30 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aditya K Kaza, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Kaza AK, Mondal A, Piekarski B, Sachse FB, Hitchcock R. Intraoperative localization of cardiac conduction tissue regions using real-time fibre-optic confocal microscopy: first in human trial. Eur J Cardiothorac Surg. 2020 Aug 1;58(2):261-268. doi: 10.1093/ejcts/ezaa040. PMID 32083653

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imaging Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imaging Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events Possibly Related to Study Intervention
Description: All adverse events will be collected and relatedness to study intervention will be determined.
Time Frame: Surgery through discharge (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Imaging Arm
Number analyzed (Participants) | 6
Participants
  Experienced AE related to study intervention | 0
  Experienced AE unrelated to study intervention | 6

2. Secondary Outcome: Number of Participants For Whom FCM Imaging During Cardiac Surgery Was Feasible
Description: Evaluated by measuring increased time on bypass, rate of enrollment, and the ability to incorporate this imaging modality into standard OR procedures. The additional time on bypass and ability to incorporate the imaging into standard OR procedures was assessed for each subject. 3 additional minutes on bypass was determined as reasonable per the protocol. The ability to incorporate the imaging was considered successful when it did not interfere with the planned clinical procedure. The rate of enrollment was evaluated for the study as a whole.
Time Frame: Surgery through discharge (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Imaging Arm
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: Percentage of Agreement in Classification of FCM Images
Description: A first reviewer selected 60 FCM images and classified them as reticulated, striated, or of poor quality (indistinguishable microstructure) with 20 images in each group. Quality of the files is measured by the ability of 8 blinded reviewers to classify the images accurately.
Time Frame: After all participants completed the study (range 2 months to 1 year post surgery)
Measure: Mean (Full Range); unit: % of agreement with unblinded reviewer
Units Other Than Participants: Images
Arm/Group | Imaging Arm
Number analyzed (Participants) | 6
Number analyzed (Images) | 60
% of agreement with unblinded reviewer | 90.4 [81.7 to 96.7]

ADVERSE EVENTS:
Time Frame: From surgery until hospital discharge, up to 9 days.
Arm/Group | Imaging Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imaging Arm (N=6)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Hypertension (Vascular disorders) | 1 (1)
Edema (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT03189134/ICF_000.pdf
  • Study Protocol (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT03189134/Prot_001.pdf